CLINICAL TRIAL: NCT07373561
Title: Post-Intensive Care Syndrome and Associated Symptom Burden Among Danish ICU Survivors: An Inception Cohort Study (PICAS-DK)
Brief Title: Post-Intensive Care Syndrome and Associated Symptom Burden Among Danish ICU Survivors
Acronym: PICAS-DK
Status: Not yet recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Camilla Bekker Mortensen, Assistant Professor, Ph.D, Critical Care Registered Nurse, Zealand University Hospital
Other Study IDs: ID not known yet
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Post-Intensive Care Syndrome (PICS); Symptom Burden; Intensive Care Unit (ICU) Patients
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: This study investigates ICU survivor patients in Denmark and aim to estimate the prevalence of post-intensive care syndrome within this group. There are three different follow-up times.

SUMMARY:
The study aims to estimate the prevalence of post-intensive care syndrome (PICS) 12 months after ICU admission among adult ICU survivors in Denmark and to describe how this prevalence is distributed across the physical, cognitive, and mental health domains. By conducting follow-up assessments at 3, 6, and 12 months post-discharge, the study further seeks to determine the prevalence of PICS at each time point, characterise its temporal trajectory, and explore patients' symptom burden over time.

Research question

* What is the prevalence of PICS and its specific components (physical, cognitive, and mental health domains) among ICU survivors 12 months after ICU admission?
* How do the components of PICS evolve during the follow-up period (trajectory)?
* What risk factors are associated with the development of PICS in ICU survivors?
* Are there differences in PICS prevalence based on demographic or clinical characteristics (e.g., age, comorbidities, ICU length of stay)?

The hypothesis is that the prevalence of post-intensive care syndrome (PICS) in a Danish cohort of adult ICU survivors at 12 months will be approximately one third, defined as impairment in at least one of the three PICS domains (physical, cognitive, or mental health), measured using validated instruments with pre-specified cut-offs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age
* Admitted to the intensive care unit for ≥48 hours
* Acutely admitted to the intensive care unit

Exclusion Criteria:

* Patients with limited treatment
* Foreign patients
* Pregnant women
* Patient with impaired cognitive function (e.g. dementia, intellectual disability)
* Patient without Danish citizenship
* Patient with limited proficiency in the Danish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish ICU-patients admitted to an intensive care unit at any of the participating hospitals in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of PICS at 12 months after ICU admission | 12 months after ICU admission
  Presence of PICS at 12 months after ICU admission, defined as impairment in at least one of the three domains (physical, cognitive or mental health) measured with validated instruments and pre-specified cut-off values.

SECONDARY OUTCOMES:
Prevalence of PICS at 3 and 6 months | Data will be collected at 3 and 6 months post-discharge
  The proportion of participants meeting the PICS definition at 3 and 6 months post-discharge, using the same domain criteria as for the 12-month primary outcome.